CLINICAL TRIAL: NCT04826380
Title: Thumb Basal Joint (CMC I) Arthritis - Preoperative Anxiety/Depression, Outcome Instruments, Carpal Kinematics and Cost-utility
Brief Title: Thumb Basal Joint (CMC I) Arthritis - Preoperative Anxiety/Depression, Outcome Instruments, Carpal Cinematics and Cost-utility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Töölö Hospital (Other)
Responsible Party: Principal Investigator, Samuli Aspinen, Principal investigator, Töölö Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3163/2020
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Arthritis; Thumb Osteoarthritis; Arthropathy; Quality of Life
MeSH Terms: conditions — Arthritis; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trapeziectomy (Other): Simple trapeziectomy for treating CMC I arthritis
  Interventions: Procedure: Trapeziectomy
- Conservative (No Intervention): Conservative measures (e.g. splint, NSAID, activation modification) for treating CMC I arthritis

INTERVENTIONS:
Procedure: Trapeziectomy — Simple trapeziectomy (without LRTI)
  Arms: Trapeziectomy

SUMMARY:
A project aiming to promote evidence based practice when treating thumb basal joint (CMC I) arthritis. We will aim to: 1) provide the minimal clinical difference of two general outcome instruments, 2) evaluate the association between pre-operative anxiety and/or depression and outcomes following trapeziectomy, 3) evaluate the effect of trapziectomy on carpal cinematics, 4) determine the cost-utility-ratio of trapeziectomy

ELIGIBILITY:
Inclusion Criteria:

* Eaton-Glickel >2 arhritis
* Symptom duration >3 months
* Pain VAS >30mm
* No significant comorbidities, ASA I-II
* Fluent in Finnish language

Exclusion Criteria:

* Eaton-Glickel <2
* Duration of symptoms <3 months
* VAS <30mm
* ASA >II
* Inflammatory joint disease
* Systemic corticosteroid or immunomodulatory medication
* Upper limb symptoms not explained with CMC I artritis
* Heavy smoking (> 20 cigarettes per day)
* Alcohol or drug abuse
* Neurological condition affecting upper limb function
* Other ipsilateral upper limb condition requiring surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist Evaluation | 12 months
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists two subscales: Pain and Function (0=best possible outcome, 10=worst possible outcome)
Michigan Hand Outcome Questionnaire | 12 months
  A hand-specific outcomes instrument that contains six distinct scales: (1) overall hand function, (2) activities of daily living, (3) pain, (4) work performance, (5) aesthetics, and (6) patient satisfaction with hand function.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | 12 months
  A pain catastrophizing scale comprising of three subscales: (1) Helplessness, (2) Rumination, and (3) Magnification
Pain (Visual Analogue Scale) | 12 months
  The VAS is derived by health care professional question of pain in scale 0 to 10 (0=no pain, 10=worst possible pain)
Global improvemen | 12 months
  Global rating to treatment effect will be evaluated by question: "How would you rate the function of your hand compared to the situation before the treatment?". The options are in 5-step Likert scale from (-2) Much worse to (+2) Much better
Grip strength | 12 months
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in kg and percentage of the unaffected side
Wrist and hand (thumb) range of motion (ROM) | 12 months
  ROM is measured on both hands with a handheld goniometer in degrees.
Cost-utility | 12 months
  Quality-adjusted life years/months measured as a change in EQ-5D
Carpal Kinematics | 12 months
  Evaluated from preoperative and compared to 1-year postoperative 4-dimension cone-beam tomography - the wrists are imaged in 7 different postures to reproduce carpal movement, the pre and postoperative scans will be compared to evalueate the effect of trapeziectomy on carpal kinematics (e.g. scapholunate angle, lunotriquetral angle, metacarpal subsidence)
Beck Depression Inventory | 12 months
  21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression

CONTACTS AND LOCATIONS:
Locations (1):
- Töölö Hospital (Helsinki University Hospital), Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analyzed during this trial will be available from the PI on reasonable request.